CLINICAL TRIAL: NCT03226054
Title: Determining Risk Factors for Successful PPI Weaning
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not logistically feasible to continue enrolling patients.
Sponsor: Mount Carmel Health System (Other)
Responsible Party: Principal Investigator, Stephanie Meller, Family Medicine Physician / Principal Investigator, Mount Carmel Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 160809-6
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Gastroesophageal Reflux
Keywords: Proton Pump Inhibitor
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Prospective Cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PPI Taper (Other): PPI Taper using Lifestyle Modifications, per study protocol
  Interventions: Behavioral: Lifestyle Modifications

INTERVENTIONS:
Behavioral: Lifestyle Modifications — Lifestyle Modifications to wean off of a Proton Pump Inhibitor, i.e. avoiding dietary triggers, waiting 3 hours to lie flat, and elevating the head of the bed

SUMMARY:
Gastroesophageal Reflux Disease ("GERD") can happen when stomach acid flows backward into your esophagus (tube from the mouth to the stomach), causing symptoms such as heartburn. Proton pump inhibitors (called "PPIs") are a type of medication that reduce acid in the stomach and are used to reduce the discomfort from GERD. Treatment for GERD with PPIs is recommended to last up to eight weeks; however, many people take them for longer periods. Some people are placed on PPIs (particularly in the hospital) to prevent ulcers and inflammation of the stomach, but they do not need to be on the medication long term. Previous research studies have shown that there are some risks with taking PPIs for a long time. These risks include the inability of your body to absorb some vitamins and minerals, certain infections such as pneumonia or the digestive tract infection called "C. diff," and possibly bone fractures. Therefore, it is desirable to stop taking a PPI when possible.

The purpose of this study is to use a standard approach to help patients stop taking PPIs by adopting lifestyle habits known to reduce the symptoms of GERD while they slowly reduce their PPI dose. All medications used for this study are approved by the U.S. Food and Drug Administration ("FDA"). You are being asked to take part in this study because you have been taking a PPI for longer than the recommended time, and have either a diagnosis of GERD, gastritis, or an unclear indication for being on a PPI. About 100 patients from the Mount Carmel St. Ann's Family Medicine practice will participate in this research.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Male or female
* PPI on home medication reconciliation
* GERD that is symptom controlled (per questionnaire), OR
* Gastritis that is symptom controlled (per questionnaire), OR
* An unclear indication for PPI use but free of GERD/gastritis/ulcer symptoms (includes patients on GI prophylaxis from the hospital and continued medication)
* Desire or willingness to be off of PPI chronically
* On PPI chronically (> 2 months or 8 weeks, can be intermittent use)
* Initial PPI dose cannot exceed more than the equivalent of Omeprazole 40mg PO BID
* Comprehend English well (per provider's discretion; to understand questionnaires, instructions, etc.)

Exclusion Criteria:

* On PPI for fewer than 2 months
* Co-morbid diagnosis of Peptic Ulcer Disease, H.pylori infection, Barrett's esophagus, malignancy, Inflammatory Bowel Disease
* Diagnosis of moderate to severe renal impairment (defined as CrCl <50 mL/min; reasoning due to caution of H2RB on renal failure)
* Diagnosis of prolonged QT interval with renal impairment (reasoning due to H2RB with concomitant renal failure may increase QT interval if not renally dosed)
* True allergy to Proton Pump Inhibitor and / or H2 Receptor Blocker
* Patients with frequent cardiac angina symptoms (decreasing the dose of PPI may cause rebound GERD and the patient may think they are having a heart attack)
* Pregnant women, fetuses, neonates or fetal material
* Females of reproductive potential at time of research that are not on a form on birth control (OCPs, tubal ligation, etc) or lactating
* Adults with decisional impairment
* Prisoners
* Patients with uncontrolled Psychological illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Successful Weaning off a Proton Pump Inhibitor | 6 months
  To eliminate GERD/gastritis symptoms and completely discontinue PPI use

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie O Meller, MD, Principal Investigator — Mount Carmel Health System
Locations (1):
- Mount Carmel St. Ann's Family Medicine Center, Westerville, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data at this time.